CLINICAL TRIAL: NCT02091570
Title: A Randomized, Controlled, Double-Blind Crossover Pilot Trial to Assess the Effects of Nutrition Bars on Subjective Ratings of Hunger and Fullness in Women
Brief Title: Effect of Nutrition Bars on Satiety in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1308
Record Dates: First submitted 2014-03-11; First posted 2014-03-19 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hunger; Satiety
Keywords: Hunger; Fullness; Satiety; Nutrition bar; Crossover

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition bar (Placebo Comparator): 50 g nutrition bar
  Interventions: Other: Nutrition Bar
- Nutrition Bar 1 (Experimental): 50 g nutrition bar with additional 2 g of milk-based nutrient
  Interventions: Other: Nutrition Bar
- Nutrition bar 2 (Experimental): 50 g nutrition bar with additional 3 g of milk-based nutrient
  Interventions: Other: Nutrition Bar

INTERVENTIONS:
Other: Nutrition Bar — Intervention involves consumption of one nutrition bar of approximately 50 g in the beginning of each visit of the crossover sequence

SUMMARY:
This study investigates nutrition bar consumption and possible impact on self-reported ratings of hunger and fullness compared to a control.

DETAILED DESCRIPTION:
Participant eligibility will be screened at visit 1. Test days will commence at 8 to 10 a.m. and visits two to four will be spaced four days apart. On visit days participants consume a nutrition bar; satiety and hunger ratings, blood samples are collected simultaneously over a three hour period. After completion, participants will complete gastrointestinal (GI) tolerability as well as Palatability and Adverse Events questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Body mass index (BMI) 20.00-29.99 kg/m2
* Maintenance of habitual diet, physical activity patterns, and body weight throughout the trial
* In general good health on the basis of medical history; and taking no medication other than birth control, hormone replacement therapy, statins or blood pressure medication
* Participant understands the study procedures, provides signed informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.
* Participant can consume a nutrition bar in the allotted time frame

Exclusion Criteria:

* Use of over-the-counter weight-loss drugs and herbal remedies or supplements and dieting programs/behavior (within two months of visit 1)
* Variation in body weight >8.8 lbs. (4 kg) within the previous three month before screening
* Any history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a health professional
* Subject scores ≥14 on restraint factor of the Three-Factor Eating Questionnaire
* History or presence of clinically important renal or gastrointestinal disorders, or diabetes mellitus
* Extreme dietary habits (e.g. vegan, Atkins diet, exclusion of major food groups, etc.)
* History of allergy, sensitivity, or strong dislike towards any of the components of the study products
* Females who are pregnant, or planning to be pregnant during the study period or lactating
* Use of an investigational drug product within the last 30 days
* Individual has a condition the Investigator believes would interfere with her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.
* Subject does not understand English.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2014-05-16 (Actual)

PRIMARY OUTCOMES:
self-reported hunger and fullness rating | 3 hour period after consumption of study product, on 3 occasions
  change in self-reported hunger or fullness compared to placebo

SECONDARY OUTCOMES:
blood sample analytes | 3 hour period after consumption of study product, on 3 occasions
  change in analyte concentrations compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Bolster, PhD, Principal Investigator — PepsiCo, Inc.; Laura Harkness, PhD, Principal Investigator — PepsiCo, Inc.
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bolster DR, Rahn M, Kamil AG, Bristol LT, Goltz SR, Leidy HJ, Blaze Mt M, Nunez MA, Guo E, Wang J, Harkness LS. Consuming Lower-Protein Nutrition Bars with Added Leucine Elicits Postprandial Changes in Appetite Sensations in Healthy Women. J Nutr. 2018 May 1;148(5):693-701. doi: 10.1093/jn/nxy023. PMID 29897544